CLINICAL TRIAL: NCT06544122
Title: Effect of Transcranial Direct Current Stimulation on the Voice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Clinical professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TDCS_voice
Record Dates: First submitted 2024-07-09; First posted 2024-08-09 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Voice and Resonance Disorders; Transcranial Direct Current Stimulation; Voice Disturbance
Keywords: transcranial direct current stimulation; voice; speech therapy
MeSH Terms: conditions — Voice Disorders; Communication Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Effects on voice of M1 tDCS in healthy voice volunteers (Active Comparator): The aim of this arm is to verify the effect on the voice of anodal tDCS M1 larynx target.
  Interventions: Device: Transcranial direct current stimulation
- Effects on voice of S1 tDCS in vocally health volunteers (Active Comparator): The aim of this arm is to verify the effect on the voice of anodal tDCS S1 larynx target.
  Interventions: Device: Transcranial direct current stimulation
- Effects on voice of PFDLC tDCS in vocally health volunteers (Active Comparator): The aim of this arm is to verify the effect on the voice of anodal tDCS PFDLC target.
  Interventions: Device: Transcranial direct current stimulation
- Effects on voice of cerebellum tDCS in vocally health volunteers (Active Comparator): The aim of this arm is to verify the effect on the voice of anodal tDCS cerebellum target.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Anodal tDCS will be applied at an intensity of 2mA and duration of 20 minutes. The assembly of the electrodes during the tDCS sessions will be carried out as follows: primary motor cortex, the stimulation electrode (anode) will be positioned on C5 (international EEG 10-20 system), in S1 (2cm posterior to C5), at the PFCDL (Fp3), all with the cathode positioned on the region contralateral supraorbital. For cerebellar tDCS the anode will be positioned on the inion area and the cathode on the deltoide muscle.
  Other Names: tDCS; transcranial electrical stimulation; anodal stimulation tDCS

SUMMARY:
The goal of this clinical trial is to verify the effect on the voice of transcranial direct current stimulation (tDCS) in vocally healthy non-singers. The main question it aims to answer is: What is the brain area in which tDCS promotes better vocal performance in vocally healthy individuals? Each participants received anodal tDCS applied at an intensity of 2 mA for a duration of 20 minutes for tDCS stimulations in different areas with a 7-day washout period between stimulations. Vocal assessments was conducted before and after the intervention. The targeted places were the primary motor cortex (M1), primary somatosensory cortex (S1), Cerebellum, and dorsolateral prefrontal cortex (DLPFC).

DETAILED DESCRIPTION:
Recently, non-invasive brain stimulation (NIBS) techniques , including transcranial direct current stimulation (tDCS), have been employed to enhance vocal skills. tDCS can be used to temporarily and reversibly modulate brain functions and is an increasingly popular tool for investigating the relationships between the brain and behavior . The aim of the present study is investigate the effect of tDCS applied to different areas on the voice of vocally healthy non-singers. This is a randomized crossover clinical trial, approved by the Research Ethics Committee of the Federal University of Pernambuco, number 5,758,856. Vocally healthy people from the city of Recife and its Metropolitan Region, aged between 18 and 45 years, participated in the study.Each participant underwent four tDCS stimulations in different areas with a 7-day washout period between stimulations to study their vocal assessments before and after tDCS. The targeted places were the primary motor cortex (M1), primary somatosensory cortex (S1), Cerebellum, and dorsolateral prefrontal cortex (DLPFC). All participants were subjected to voice acessments analysis immediately before and after tDCS application in each area. Data normality will be analyzed using the Shapiro-Wilk test, rejecting the hypothesis of normal distribution when p<0.05. ANOVA will be applied to design repeated measures in case of normality and in the existence of asymmetric data, Friedmann's ANOVA will be used for repeated measures. For the comparison of values before and after application of the technique and between modes of execution of the technique (with and without non-invasive neuromodulation), tests will be applied for related and independent samples, respectively, with a significance level of 5%

ELIGIBILITY:
Inclusion Criteria:

* Non-singers with healthy voice

Exclusion Criteria:

* Smokers
* Those who present signs and symptoms of laryngeal, pharyngeal or respiratory diseases at the time of collection
* Volunteers who make regular use of neuroactive drugs
* Those who have metallic implants or a pacemaker
* People that have any history of seizures or epilepsy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
Vocal range profile | through study completion, an average of 6 months
  Min f0 (Hz) Max f0 (Hz) Ext f0 (Hz) Ext (ST) Mín int (dB) Max int (dB) Area (%)
  Min f0 (Hz) Max f0 (Hz) Ext f0 (Hz) Ext (ST) Mín int (dB) Max int (dB) Area (%)
  Minimum f0 (Hz); Maximum f0 (Hz); Extension f0; Extension in St; Minimum intensity (dB); Maximum intensity (dB); Area (%)

SECONDARY OUTCOMES:
Voice | through study completion, an average of 6 months
  Jitter (%); Shimmer (%); Irregularity; GNE; DAI
Laryngeal diadochokinesis | through study completion, an average of 6 months
  Change in the task of producing vowels separately, with rapid repetition of each vowel as quickly as possible for eight seconds
Vocal effort | through study completion, an average of 6 months
  The Adapted Borg CR10 for Vocal Effort Ratings (BR) maintained a scale from 0 to 10, where 0 means "no vocal effort at all", and 10 "maximum vocal effort". First, the participants have to reproduce a note played on a virtual keyboard (3 tones below their maximum glissando frequency) and sustain the note while counting from 21 to 30, immediately afterwards, the participants answered the Adapted Borg CR10 for Vocal Effort Ratings (BR).

CONTACTS AND LOCATIONS:
Overall Officials: kelly Greyce SC Oliveira, PhD student, Principal Investigator — UFPE
Locations (1):
- Laboratório de Neurociência Aplicada, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Behroozmand R, Johari K, Bridwell K, Hayden C, Fahey D, den Ouden DB. Modulation of vocal pitch control through high-definition transcranial direct current stimulation of the left ventral motor cortex. Exp Brain Res. 2020 Jun;238(6):1525-1535. doi: 10.1007/s00221-020-05832-9. Epub 2020 May 23. PMID 32447409
- [Background] Peng D, Lin Q, Chang Y, Jones JA, Jia G, Chen X, Liu P, Liu H. A Causal Role of the Cerebellum in Auditory Feedback Control of Vocal Production. Cerebellum. 2021 Aug;20(4):584-595. doi: 10.1007/s12311-021-01230-1. Epub 2021 Feb 8. PMID 33555544
- [Background] Thair H, Holloway AL, Newport R, Smith AD. Transcranial Direct Current Stimulation (tDCS): A Beginner's Guide for Design and Implementation. Front Neurosci. 2017 Nov 22;11:641. doi: 10.3389/fnins.2017.00641. eCollection 2017. PMID 29213226
- [Background] Wang B, Xiao S, Yu C, Zhou J, Fu W. Effects of Transcranial Direct Current Stimulation Combined With Physical Training on the Excitability of the Motor Cortex, Physical Performance, and Motor Learning: A Systematic Review. Front Neurosci. 2021 Apr 9;15:648354. doi: 10.3389/fnins.2021.648354. eCollection 2021. PMID 33897361
- [Background] Perikova E, Blagovechtchenski E, Filippova M, Shcherbakova O, Kirsanov A, Shtyrov Y. Anodal tDCS over Broca's area improves fast mapping and explicit encoding of novel vocabulary. Neuropsychologia. 2022 Apr 15;168:108156. doi: 10.1016/j.neuropsychologia.2022.108156. Epub 2022 Jan 10. PMID 35026217
- [Background] Cardoso NSV, Lucena JA, de Lira ZS, de Vasconcelos SJ, Lopes LW, Gomes AOC. Do Flexible Silicone Tubes Immersed in Water Combined With Vocalise Improve the Immediate Effect on Voice? J Speech Lang Hear Res. 2021 Dec 13;64(12):4535-4562. doi: 10.1044/2021_JSLHR-20-00629. Epub 2021 Nov 11. PMID 34762812
- See also: Immediate Effect of a Resonance Tube on the Vocal Range Profile of Choristers — https://doi.org/10.1016/j.jvoice.2019.01.006

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT06544122/Prot_SAP_000.pdf